CLINICAL TRIAL: NCT02318953
Title: The Effect of Mobile App Home Monitoring on the Number of In-Person Visits Following Ambulatory Surgery: A Randomized Control Trial
Brief Title: The Effect of Mobile App Home Monitoring on the Number of In-Person Visits Following Ambulatory Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013 0094 B
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Use of Mobile App Home Monitoring After Ambulatory Surgery
Keywords: Telemedicine; Ambulatory Surgical Procedures; Postoperative Care; Cost Effectiveness; Mobile Applications; Health Services Research; Breast Reconstruction
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile app follow-up care (Experimental): The mobile app follow-up group will have no planned in-person follow-up at one- and four weeks postoperative. However, these visits will be replaced with surgical site examination via submitted photos, visual analog scale (VAS) to assess pain, and the quality of recovery-9 (QoR9) questionnaire monitoring. All of this information is submitted via the mobile application (QoC Health Inc. Toronto). Patient will use daily monitoring for two weeks and then weekly monitoring for four weeks. The surgeon will use a wireless interface to access that data and monitor the patient's condition (not in real time). Physicians will summarize the clinical findings recorded by the mobile app at one week and four weeks postoperative using the prototypical "SOAP" note.
  Interventions: Device: Mobile app follow-up care
- Conventional, in-person follow-up care (Active Comparator): Patients in the conventional, in-person follow-up group will have a planned clinic follow-up at one- and 4-weeks postoperative. This is the follow-up schedule currently used by both surgeons. At these scheduled follow-ups, patients will be asked to complete the VAS to assess pain and the QoR9 questionnaire.
  Interventions: Other: Conventional, in-person follow-up care

INTERVENTIONS:
Device: Mobile app follow-up care — The mobile app follow-up care is an application that can be loaded on to a smartphone. It allows the patient to submit photos of their surgical site, VAS pain scores, and QoR9 scores. The information collected is transmitted to members of the surgical team (i.e. the primary surgeon) and used to monitor recovery over the first 30-days following surgery.
  Other Names: QoC Health Inc. mobile application
  Arms: Mobile app follow-up care
Other: Conventional, in-person follow-up care — This includes a typical in-person visit with the operating surgeon at one- and four-weeks after surgery.
  Arms: Conventional, in-person follow-up care

SUMMARY:
This study evaluate if in an ambulatory breast reconstruction patient population at Women's College Hospital (WCH), can we avert in-person follow-up care through the use of mobile app home monitoring compared to conventional, in-person follow-up care in the first 30-days following surgery.

DETAILED DESCRIPTION:
Women's College Hospital offers specialized surgical procedures, including breast reconstruction. Patients often travel great distances to undergo surgery. The average ambulatory breast reconstruction patient travels 76 km from home to hospital, with the furthest patient coming from 540 km away.

Most patients receiving ambulatory breast reconstruction have a low rate of postoperative events necessitating clinic visits. However, regular follow-up is still considered important in the early post-operative phase. Increasingly, telemedicine is used to overcome the distance patients must travel to receive specialized care. Telemedicine data suggests that mobile monitoring and follow-up care is valued by patients and can reduce costs to society (1-3).

Currently, Women's College Hospital is using a mobile application (QoC Health Inc., Toronto) to complement in-person postoperative follow-up care for breast reconstruction patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing breast reconstruction at Women's College Hospital. They must be able to use a mobile device and communicate in English.

Exclusion Criteria:

* They must be non-smokers because smokers carry increased rates of complication and both surgeons have a policy to solely operate on non-smokers (minimum smoke-free period of one month leading to surgery). Pain ratings captured in the VAS and QoR9 are important for judging quality of postoperative recovery. Pre-existing pain or an inability to take narcotics would compromise the reliability of these measures. Therefore, patients must not suffer from chronic pain. They must not be taking narcotic (morphine-like) medication for pain on a regular basis. They must not have an allergy to local anesthetics or morphine-like medications.

Accommodation of special populations: Patients with hearing or speaking impairments will be accommodated with the help of translator. The person who regularly attends visits with her will facilitate this, or if no such person is available, we will use a hospital translator. All patients will receive an explanation of the study and the consent form in writing. All material will be understandable by patients with a grade 6 reading level. If our patients have lower than a grade 6 reading level, we will ask them if there is a family member at home who could assist them with the use of the mobile device.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The total number of physician visits related to the surgery | 30 days
  The total number of physician visits will include visits to the specialist, family physician, and emergency department related to surgery. This data will be captured by patient survey at two- and four-weeks after surgery.

SECONDARY OUTCOMES:
The total number of health care telephone calls and emails related to the surgery. | 30 days
  The total number of health care telephone calls and emails will include specialist, family physician, and emergency services. This data will be captured by patient survey at two- and four-weeks after surgery.
Number of complications | 30 days
  We will record and report all complications occurring within the 30-day period. This was chosen based on literature surrounding postoperative complications in the first 30-days (4). This will be captured by patient survey at two- and four-weeks after surgery.
Societal and healthcare system costs | 30 days
  A societal perspective will be adopted wherein all cost are assessed irrespective of the payer. This perspective was chosen based on the US Panel on Cost-Effectiveness in Health and Medicine recommendations. This recommendation is meant to improve comparability and consistency across studies (5). Furthermore, while a broad societal perspective will be adopted, results will also be presented using a narrower health system perspective that may be of key interest to health administrators and policy decision makers. This alternative perspective focuses on costs borne within the health system and excludes external costs as well as costs borne by patients and their caregivers.
Patient satisfaction | 30 days
  Currently, there are no validated questionnaires that capture patient satisfaction with postoperative care. We have created a post-pilot survey that captures patient satisfaction with the care and information received. All answers are recorded using a 5-point likert scale. This will be captured at four-weeks after surgery. We will also use the QoR-9 scores and pain VAS scores recorded at one- and four-weeks postoperative. Psychometric properties of the QoR9 include convergent validity and discriminant construct validity. There is also good interrater agreement and internal consistency. The test-retest reliability was 0.61 (p<0.0001). The preferred cut-off is 0.7; however, the QoR9 was still favoured over the quality of recovery-40 (QoR40) questionnaire due to its ease of use (< 2 minutes required to complete the survey) (6). This will be captured in both groups at one- and four-weeks after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: John Semple, MD, MSc, Principal Investigator — University of Toronto
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hwa K, Wren SM. Telehealth follow-up in lieu of postoperative clinic visit for ambulatory surgery: results of a pilot program. JAMA Surg. 2013 Sep;148(9):823-7. doi: 10.1001/jamasurg.2013.2672. PMID 23842982
- [Background] Jones DT, Yoon MJ, Licameli G. Effectiveness of postoperative follow-up telephone interviews for patients who underwent adenotonsillectomy: a retrospective study. Arch Otolaryngol Head Neck Surg. 2007 Nov;133(11):1091-5. doi: 10.1001/archotol.133.11.1091. PMID 18025311
- [Background] Bailey J, Roland M, Roberts C. Is follow up by specialists routinely needed after elective surgery? A controlled trial. J Epidemiol Community Health. 1999 Feb;53(2):118-24. doi: 10.1136/jech.53.2.118. PMID 10396473
- [Background] Kazaure HS, Roman SA, Sosa JA. Association of postdischarge complications with reoperation and mortality in general surgery. Arch Surg. 2012 Nov;147(11):1000-7. doi: 10.1001/2013.jamasurg.114. PMID 23165614
- [Background] Siegel JE, Weinstein MC, Russell LB, Gold MR. Recommendations for reporting cost-effectiveness analyses. Panel on Cost-Effectiveness in Health and Medicine. JAMA. 1996 Oct 23-30;276(16):1339-41. doi: 10.1001/jama.276.16.1339. PMID 8861994
- [Background] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071
- [Derived] Armstrong KA, Coyte PC, Brown M, Beber B, Semple JL. Effect of Home Monitoring via Mobile App on the Number of In-Person Visits Following Ambulatory Surgery: A Randomized Clinical Trial. JAMA Surg. 2017 Jul 1;152(7):622-627. doi: 10.1001/jamasurg.2017.0111. PMID 28329223
- [Derived] Armstrong KA, Coyte PC, Bhatia RS, Semple JL. The effect of mobile app home monitoring on number of in-person visits following ambulatory surgery: protocol for a randomized controlled trial. JMIR Res Protoc. 2015 Jun 3;4(2):e65. doi: 10.2196/resprot.4352. PMID 26040252